CLINICAL TRIAL: NCT05656365
Title: Evaluating the Genetics and Immunology of Periodic Fever, Aphthous Stomatitis, Pharyngitis, and Cervical Adenitis (PFAPA) Syndrome and Other Tonsil Disorders
Status: Recruiting | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10001043; 001043-I
Record Dates: First submitted 2022-12-15; First posted 2022-12-19 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11-13

CONDITIONS: Periodic Fever, Aphthous Stomatitis, Pharyngitis, And Cervical Adenitis (Pfapa); Obstructive Sleep Apnea; Tonsillitis; Tonsil Disorder; Sleep Disordered Breathing
Keywords: Genome-Wide Association Study (Gwas); Immunology; Autoinflammation; Tonsillitis; Obstructive Sleep Apnea; Sleep Disordered Breathing; Natural History
MeSH Terms: conditions — Hereditary Autoinflammatory Diseases; Stomatitis, Aphthous; Pharyngitis; Sleep Apnea, Obstructive; Tonsillitis; Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Patients with periodic fever, aphthous stomatitis, pharyngitis, and cervical adenitis (PFAPA) syndrome and other tonsil disorders.

SUMMARY:
Background:

Periodic fever, aphthous stomatitis, pharyngitis, and cervical adenitis (PFAPA) is the most common periodic fever syndrome of childhood. Symptoms can include swelling of the glands in the throat, mouth ulcers, and tonsillitis. Removal of the tonsils can stop the periodic flareups. But researchers do not know how PFAPA develops. In this natural history study, researchers will collect specimens and data from people with PFAPA to see what they might have in common.

Objective:

To collect blood and other specimens from people with PFAPA to learn more about the illness.

Eligibility:

People aged 1 month or older with symptoms of PFAPA or another tonsil disorder.

Design:

Participants will be screened. Their medical records will be reviewed. Researchers will ask about a family history of PFAPA.

The following specimens may be collected:

Blood. Blood will be drawn either from a needle inserted into a vein or from a prick in the finger or heel.

Mucus and cells. A stick with soft padding on the tip may be rubbed inside the nostrils or mouth.

Stool.

Saliva.

Tissue samples may be taken if participants are having surgery to remove the tonsils or adenoids. Participants having surgery may also have a nasopharyngeal wash; salt water will be squirted into the back of the throat and then sucked back out with a syringe.

Most participants will provide specimens only once. They can do this in person at the clinic; they can also have their local health providers send specimens to the researchers. Some participants may have optional follow-up visits over 10 years.

DETAILED DESCRIPTION:
Study Description:

The purpose of this multisite study is to collect specimens and data from patients with periodic fever, aphthous stomatitis, pharyngitis, and cervical adenitis (PFAPA) syndrome and other tonsil disorders for genetic, immunologic, cellular, molecular, and microbial research into the pathogenesis of these conditions. Specimens include blood, saliva, buccal swabs, oropharyngeal swabs, nasopharyngeal swabs, nasopharyngeal wash, and/or stool. If a participant is scheduled to undergo a clinically indicated tonsillectomy and/or adenoidectomy, then leftover clinical specimens will also be collected for research. Participants may either be seen in person at the study sites or may be seen remotely via telehealth and provide send-in samples collected locally.

Primary Objective:

To collect samples to understand the immunologic mechanisms and genetic and microbial risk factors for PFAPA and other tonsil disorders.

Primary Endpoints:

1. Identify genetic risk variants for PFAPA and other tonsil disorders.
2. Characterize immune cell populations, gene expression (including at the single-cell level), epigenetic features, and protein expression ex vivo in blood, tissue, washes, or swabs from people with PFAPA and other tonsil disorders.
3. Characterize the tonsillar/adenoid, oral, nasal and/or stool microbiota in people with PFAPA and other tonsil disorders.
4. Characterize clinical outcomes following tonsillectomy and other clinically indicated treatments.

Secondary Objective: To understand the characteristics and function of unique cell populations in the pharyngeal lymphoid tissues (tonsils and adenoids) and how immune responses to antigens are generated in these tissues.

Secondary Endpoints:

1. Study responses to antigens and infection in the mucosal lymphoid tissue and peripheral blood.
2. Characterize unique immune cell populations present in the mucosal tissue.
3. Characterize immunologic and molecular pathways in the tissue cells.

ELIGIBILITY:
* INCLUSION CRITERIA:

Participants must meet all the following inclusion criteria to be eligible for this study:

1. Aged >=1 month. To be seen at the NIH CC, participants must be >=3 years of age.
2. Diagnosed with PFAPA or another tonsil disorder, or has symptoms consistent with these conditions, as determined by the investigator.
3. Able to provide informed consent (for ages >=18 years) or has a parent or guardian who can provide informed consent on their behalf (for ages <18 years).
4. Willing to allow specimens and data to be stored for future research.
5. Willing to allow genetic testing on their biospecimens.

EXCLUSION CRITERIA:

An individual who has any condition that, in the judgment of the investigator, may put them at undue risk or make them unsuitable for participation in the study will be excluded.

Ages: 1 Month to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with PFAPA and other tonsil disorders.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2023-05-23 (Actual); Primary Completion 2037-06-30 (Estimated); Study Completion 2038-12-31 (Estimated)

PRIMARY OUTCOMES:
Identify genetic risk variants for PFAPA and other tonsil disorders | Throughout study
  To collect samples to understand the immunologic mechanisms and genetic and microbial risk factors for PFAPA and other tonsil disorders
Characterize clinical outcomes following tonsillectomy and other clinically indicated treatments. | Throughout study
  To collect samples to understand the immunologic mechanisms and genetic and microbial risk factors for PFAPA and other tonsil disorders
Characterize the tonsillar/adenoid, oral, nasal and/or stool microbiota in people with PFAPA and other tonsil disorders | Throughout study
  To collect samples to understand the immunologic mechanisms and genetic and microbial risk factors for PFAPA and other tonsil disorders
Characterize immune cell populations, gene expression including at the single cell level, epigenetic features, and protein expression ex vivo in blood, tissue, washes, or swabs from people with PFAPA and other tonsil disorders | Throughout study
  To collect samples to understand the immunologic mechanisms and genetic and microbial risk factors for PFAPA and other tonsil disorders

SECONDARY OUTCOMES:
Characterize immunologic and molecular pathways in the tissue cells. | Throughout study
  To understand the characteristics and function of unique cell populations in the pharyngeal lymphoid tissues (tonsils and adenoids) and how immune responses to antigens are generated in these tissues
Study responses to antigens and infection in the mucosal lymphoid tissue and peripheral blood. | Throughout study
  To understand the characteristics and function of unique cell populations in the pharyngeal lymphoid tissues(tonsils and adenoids) and how immune responses to antigens are generated in these tissues
Characterize unique cell populations and the immunologic and molecular pathways in the tissue cells | Throughout study
  To understand the characteristics and function of unique cell populations in the pharyngeal lymphoid tissues (tonsils and adenoids) and how immune responses to antigens are generated in these tissues

CONTACTS AND LOCATIONS:
Overall Officials: Kalpana Manthiram, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (3):
- United States (3):
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Indiana University School of Medicine, Indianapolis, Indiana
  - National Institutes of Health Clinical Center, Bethesda, Maryland

IPD SHARING:
Plan to Share IPD: Yes
Deidentified IPD that underlie results in a publication or associated with genomic data deposited in a data base will be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Will be shared at the time of publication or data deposition into data base.
Access Criteria: Individual level data in dbGaP is controlled access as investigators must place a request and be approved by dbGaP. Aggregated data will be open access.

REFERENCES:
- [Background] Xu Q, Milanez-Almeida P, Martins AJ, Radtke AJ, Hoehn KB, Oguz C, Chen J, Liu C, Tang J, Grubbs G, Stein S, Ramelli S, Kabat J, Behzadpour H, Karkanitsa M, Spathies J, Kalish H, Kardava L, Kirby M, Cheung F, Preite S, Duncker PC, Kitakule MM, Romero N, Preciado D, Gitman L, Koroleva G, Smith G, Shaffer A, McBain IT, McGuire PJ, Pittaluga S, Germain RN, Apps R, Schwartz DM, Sadtler K, Moir S, Chertow DS, Kleinstein SH, Khurana S, Tsang JS, Mudd P, Schwartzberg PL, Manthiram K. Adaptive immune responses to SARS-CoV-2 persist in the pharyngeal lymphoid tissue of children. Nat Immunol. 2023 Jan;24(1):186-199. doi: 10.1038/s41590-022-01367-z. Epub 2022 Dec 19. PMID 36536106
- [Background] Manthiram K, Preite S, Dedeoglu F, Demir S, Ozen S, Edwards KM, Lapidus S, Katz AE; Genomic Ascertainment Cohort; Feder HM Jr, Lawton M, Licameli GR, Wright PF, Le J, Barron KS, Ombrello AK, Barham B, Romeo T, Jones A, Srinivasalu H, Mudd PA, DeBiasi RL, Gul A, Marshall GS, Jones OY, Chandrasekharappa SC, Stepanovskiy Y, Ferguson PJ, Schwartzberg PL, Remmers EF, Kastner DL. Common genetic susceptibility loci link PFAPA syndrome, Behcet's disease, and recurrent aphthous stomatitis. Proc Natl Acad Sci U S A. 2020 Jun 23;117(25):14405-14411. doi: 10.1073/pnas.2002051117. Epub 2020 Jun 9. PMID 32518111
- [Background] Stojanov S, Lapidus S, Chitkara P, Feder H, Salazar JC, Fleisher TA, Brown MR, Edwards KM, Ward MM, Colbert RA, Sun HW, Wood GM, Barham BK, Jones A, Aksentijevich I, Goldbach-Mansky R, Athreya B, Barron KS, Kastner DL. Periodic fever, aphthous stomatitis, pharyngitis, and adenitis (PFAPA) is a disorder of innate immunity and Th1 activation responsive to IL-1 blockade. Proc Natl Acad Sci U S A. 2011 Apr 26;108(17):7148-53. doi: 10.1073/pnas.1103681108. Epub 2011 Apr 8. PMID 21478439
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001043-I.html